CLINICAL TRIAL: NCT02820454
Title: Etude Clinique de Phase I de Radiosensibilisation de métastases cérébrales Par Nanoparticules de Gadolinium
Brief Title: Radiosensitization of Multiple Brain Metastases Using AGuIX Gadolinium Based Nanoparticles
Acronym: NANO-RAD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: NH TherAguix SAS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC15.278; 2015-004259-30 (EudraCT Number)
Record Dates: First submitted 2016-06-02; First posted 2016-07-01 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-04

CONDITIONS: Brain Metastases
Keywords: AGuIX; polysiloxane gadolinium-chelates based nanoparticles
MeSH Terms: conditions — Brain Neoplasms | interventions — AGuIX

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AGuIX and radiotherapy (Experimental): Patients receive a single intravenous injection of AGuIX on day 1. Then patients undergo a whole brain radiation therapy, 5 days a week in weeks 1-2. The first radiotherapy session will be performed 4 hours after AGuIX injection.
  Five dose escalation cohorts : 15 mg/kg, 30mg/kg, 50mg/kg, 75mg/kg and 100 mg/kg
  Interventions: Drug: AGuIX; Radiation: whole brain radiation therapy

INTERVENTIONS:
Drug: AGuIX — A single intravenous injection on day 1. Dose level 1: 15mg/kg; Dose level 2: 30mg/kg, Dose level 3: 50mg/kg; Dose level 4: 75mg/kg; Dose level 5: 100mg/kg
  Other Names: Nano-sized gadolinium particles
Radiation: whole brain radiation therapy — 30Gy in 10 sessions of 3Gy (5 days a week in weeks 1-2); first session 4 hours after AGuIX injection.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. AGuIX particles may increase the effectiveness of radiation therapy by making tumor cells more sensitive to radiation.

PURPOSE: This first-in-man Phase I trial will study the side effects and best dose of AGuIX when injected together with whole brain radiation therapy in treating patients with multiple brain metastases. The effectiveness of the combination of AGuIX and radiation therapy will be also assessed.

DETAILED DESCRIPTION:
The present study will investigate the safety, tolerability and spectrum of side effects of AGuIX in combination with whole brain radiation therapy. As such, this study will characterize the dose limiting toxicities (DLT) and maximum tolerated dose (MTD) of in combination with whole brain radiation therapy in patients with multiple brain metastases.

On day 1, patients will receive a single intravenous injection of AGuIX. An MRI scan will be performed 2 hours after injection to visualize the distribution of AGuIX in brain metastases and surrounding healthy tissue, and to evaluate the contrast enhancement in brain metastases. Then patients will undergo a whole brain radiation therapy, starting 4 hours after AGuIX injection, up to completion of 2 weeks, 5 days a week of treatment (30Gy, 3Gy/fraction).

During the first 24h after injection, several blood draws will be also performed in order to assess the pharmacokinetic of AGuIX.

After completion of study treatment, patients will be followed periodically.

Patients will be enrolled in cohorts and will be treated at sequentially rising dose levels of AGuIX combined with whole brain radiation therapy. Three subjects will initially enter at each dose. If none of the three experiences a dose-limiting toxicity we will proceed to the next dose. If one of the three experiences that level of toxicity, we will accrue 3 more subjects at that dose. If at any time there are two or more dose-limiting toxicities (in the 3-6 subjects) on a given dose, we will drop down to a lower dose. Dose escalation will continue until the MTD of AGuIX and whole brain radiation therapy is established. The MTD will then be one dose below the DLT occurring in at least 1 out of 3 subjects (2 out of 6 patients).

ELIGIBILITY:
Inclusion criteria:

* Patients with brain metastasis ineligible for local treatment by surgery or stereotactic radiation
* At least 18 years old
* Secondary brain metastases from a histologically confirmed solid tumor
* Patient competent to give informed consent (ou Signed informed consent after informing the patient)
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 3
* No prior brain irradiation
* No renal insufficiency (glomerular filtration rate > 60 mL/min/1.73m²)
* Normal liver function (bilirubin < 30 µmol/L; Alkaline phosphatase < 400 UI/L; Aspartate aminotransferase (AST) < 75 UI/L; Alanine aminotransferase (ALT) < 175 UI/L)
* For both male and female patients, effective methods of contraception must be used throughout the study. Acceptable methods of contraception are oral or implantable contraceptives, intrauterine device, condoms, spermicidal gels, or surgical sterilization.
* Affiliated to a social security scheme or assimilated

Exclusion criteria:

* Meningeal carcinomatosis
* Progressive and threatening extracranial disease
* Previous cranial irradiation (whether whole or partial brain radiation therapy, except stereotactic irradiation) or total body irradiation
* Known contra-indication, sensitivity or allergy to gadolinium
* Patients unable to undergo or tolerate Magnetic Resonance Imaging
* Patients participating in another clinical investigation at the time
* Protected persons under articles L1121-5 to L1121-8, Code of Public Health

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Maximum-tolerated dose (MTD) of polysiloxane gadolinium-chelates based nanoparticles (AGuIX) given concurrently to the whole brain radiation therapy for the treatment of multiple brain metastases | 18 months
  To determine Maximum-tolerated dose (MTD) of polysiloxane gadolinium-chelates based nanoparticles (AGuIX) given concurrently to the whole brain radiation therapy, according to incidence of dose limiting toxicity (DLT) graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03

SECONDARY OUTCOMES:
Pharmacokinetic characteristics of AGuIX particles after intravenous injection | 18 months
  Cmax
Pharmacokinetic characteristics of AGuIX particles after intravenous injection | 18 months
  AUC
Pharmacokinetic characteristics of AGuIX particles after intravenous injection | 18 months
  T1/2
Distribution of AGuIX particles in brain metastases and surrounding healthy tissue evaluated by MRI | 30 months
  Measure of the T1 contrast enhancement in brain metastases and surrounding healthy tissue after intravenous administration of AGuIX particles
Intracranial progression-free survival | 12 months after radiation
  The intracranial progression-free survival will be assessed by MRI (1,3, 6, 9 and 12 months from the date of discovery of the metastases)
Overall survival | 30 months
  The overall survival will be assessed starting from the date of discovery of the metastases

CONTACTS AND LOCATIONS:
Overall Officials: Camille VERRY, MD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Verry C, Sancey L, Dufort S, Le Duc G, Mendoza C, Lux F, Grand S, Arnaud J, Quesada JL, Villa J, Tillement O, Balosso J. Treatment of multiple brain metastases using gadolinium nanoparticles and radiotherapy: NANO-RAD, a phase I study protocol. BMJ Open. 2019 Feb 11;9(2):e023591. doi: 10.1136/bmjopen-2018-023591. PMID 30755445